CLINICAL TRIAL: NCT02995655
Title: A Pilot Study of CX-01 Combined With Azacitidine in the Treatment of Relapsed or Refractory Myelodysplastic Syndrome and Acute Myeloid Leukemia
Brief Title: CX-01 Combined With Azacitidine in the Treatment of Relapsed or Refractory Myelodysplastic Syndrome and Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Cantex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201608032; CNTX-CX-01-2016-MDS-1 (Other: Cantex Pharmaceuticals)
Record Dates: First submitted 2016-12-13; First posted 2016-12-16 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia; AML; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — N-desulfated,2-O,3-O-desulfated heparin; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CX-01 + Azacitidine (Experimental): * CX-01 will be administered as a 5-minute bolus infusion at a dose of 4mg/kg on Day 1 of each 28-day cycle, followed by a continuous intravenous infusion at a dose of 0.25 mg/kg/hour for Days 1 through 7 of each cycle. The dose of CX-01 should be calculated based on actual body weight (kg) as measured on Day 1 of each cycle.
  * Azacitidine will be administered as a 15-minute intravenous infusion at a dose of 75mg/m^2 on Days 1-7 of each 28-day cycle. Azacitidine dose should be calculated based on actual body weight and height to determine BSA. CX-01 may be administered before or after azacitidine, at the discretion of the treating physician.
  * Up to 6 cycles of treatment allowed
  Interventions: Drug: CX-01; Drug: Azacitidine; Procedure: Bone marrow biopsy; Procedure: Peripheral blood draw

INTERVENTIONS:
Drug: CX-01 — CX-01 at a dose of 4mg/kg on Day 1 of each 28-day cycle, followed by a continuous intravenous infusion at a dose of 0.25 mg/kg/hour for Days 1 through 7 of each cycle.
  Other Names: 2-O, 3-O desulfated heparin; ODSH
Drug: Azacitidine — Azacitidine at a dose of 75mg/m^2 on Days 1-7 of each 28-day cycle.
  Other Names: Vidaza®; Ladakamycin
Procedure: Bone marrow biopsy — -Baseline, day 28 of even-numbered cycle through Cycle 6, and end of study
Procedure: Peripheral blood draw — -Day 1 of each cycle, day 3 of each cycle, day 7 of each cycle, day 28 of every even-numbered cycle through Cycle 6, and end of study

SUMMARY:
The investigators hypothesize that CX-01 will disrupt the bone marrow microenvironment and increase the cytotoxic effects of azacitidine on myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML) hematopoietic stem cells by disrupting the High-mobility group box protein 1 (HMGB1) interaction with toll-like receptor 4 (TLR4) and receptors for advanced glycation end products (RAGE), the CXC chemokine CXCL12/chemokine receptor 4 (CXCR4) axis, and by disrupting other leukocyte and vascular adhesion molecules. In addition, CX-01 may also help promote count recovery after treatment given its affinity for platelet factor-4 (PF4).

The selection of CX-01 dose for study in relapsed or refractory MDS and AML has been based upon the dual requirements to have sufficient drug administered to have potential activity but without clinically significant anticoagulation. The study dose chosen (4 mg/kg bolus followed by 0.25 mg/kg/hour) fulfills both of these criteria. In addition, this dose is expected to result in serum levels of CX-01 which are significantly higher than the IC90 identified in preclinical studies for inhibition of HMGB1-RAGE, toll-like receptor 2 (TLR2) and TLR4 interaction. Therefore, the chosen dose represents a rational balance between effective dosing and safety in thrombocytopenic patients with MDS and AML. This dose was previously established to be safe and tolerable when combined with cytarabine and idarubicin in patients with AML.

ELIGIBILITY:
Inclusion Criteria:

* One of the following diagnoses:

  * MDS with International Prostate Symptom Score (IPSS) score of INT-1 or higher and one of the following:

    * Symptomatic anemia with either hemoglobin < 10.0 g/dL or requiring red blood cell (RBC) transfusion
    * Thrombocytopenia with a history of two or more platelet counts < 50,000/µL or a significant hemorrhage requiring platelet transfusions
    * Neutropenia with two or more absolute neutrophil count (ANC) < 1,000/µL
  * Non-M3 AML
* Prior treatment with ≥ 4 cycles of a hypomethylating agent (decitabine or azacitidine) without response OR documented disease progression on or after hypomethylating agent therapy
* Age ≥ 18 years old
* Adequate renal and hepatic function defined as all of the following:

  * total bilirubin ≤ 1.5 x upper limit of normal (ULN), except in cases of Gilbert's disease
  * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
  * serum creatinine < 2.0 x ULN
* Peripheral blood blast count < 10,000/ µL.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Females must be surgically or biologically sterile or postmenopausal or, if of childbearing potential, must agree to use an adequate method of contraception during the study until 30 days after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 30 days after the last treatment.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior allogeneic stem cell transplant
* Central nervous system (CNS) leukemia
* Diagnosed with AML and eligible for standard induction chemotherapy or stem cell transplantation.
* At an increased risk of hemorrhage.
* Known allergies, hypersensitivity, or intolerance to any form of heparin or azacitidine
* Presence of significant active bleeding or condition requiring maintenance of a platelet count > 50,000/µL
* Presence of any condition requiring any form of anticoagulant therapy (heparin flushes for IV catheter are permitted)
* Receiving concomitant chemotherapy, radiation therapy, or immunotherapy during the duration of treatment on protocol, or within 21 days prior to enrollment
* Known seropositivity for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 28 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Overall response rate (partial response or higher) | 30 days following completion of treatment (estimated to be 28 weeks)
  * Overall response rate = the percentage of patients obtaining partial response or higher
  * Patients will be assessed for response according to modified International Working Group (IWG) criteria

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 5 years
  * The interval from the date of first dose of study drug to disease progression or death.
  * Described by median time-to-event and a 95% confidence interval, if estimable, using Kaplan-Meier models
Disease-free survival (DFS) | Up to 5 years
  * The interval from the date of first documentation of a CR to date of recurrence or death. This is determined only for patients achieving a CR
  * Described by median time-to-event and a 95% confidence interval, if estimable, using Kaplan-Meier models
Overall survival (OS) | Up to 5 years
  * The date of first dose of study drug to the date of death from any cause.
  * Described by median time-to-event and a 95% confidence interval, if estimable, using Kaplan-Meier models
Safety and tolerability of regimen as measured by adverse events tabulated by patient | 30 days following completion of therapy (estimated to be 28 weeks)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 will be utilized for all toxicity reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Westervelt, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu